CLINICAL TRIAL: NCT04581473
Title: An Open, Multicenter, Phase Ib/II Study to Evaluate the Efficacy, Safety and Pharmacokinetics of CT041 Autologous CAR T-cell Injection in Patients With Advanced Gastric/ Gastroesophageal Junction Adenocarcinoma and Pancreatic Cancer
Brief Title: Study to Evaluate the Efficacy, Safety and Pharmacokinetics of CT041 Autologous CAR T-cell Injection
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Collaborators: Peking University Cancer Hospital & Institute (Other); Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT041-ST-01
Record Dates: First submitted 2020-09-24; First posted 2020-10-09 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Gastric Adenocarcinoma; Pancreatic Cancer; Gastroesophageal Junction Adenocarcinoma
Keywords: advanced solid tumors; Gastric Cancer; Pancreatic Cancer; Esophagogastric Junction Cancer; Claudin18.2; CLDN18.2; CAR T cell
MeSH Terms: conditions — Pancreatic Neoplasms; Stomach Neoplasms | interventions — Immunotherapy, Adoptive; Irinotecan; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CT041 autologous CAR T-cell injection (Experimental): Two stages: Phase 1b: dose escalation and dose expansion; Phase 2: verify CT041 efficacy and safety
  Interventions: Drug: CT041 autologous CAR T-cell injection
- Physician's Choice (Active Comparator): Participants will receive physician's choice of treatment in Phase II
  Interventions: Drug: Physician's Choice（Paclitaxel or Irinotecan or Apatinib or Anti-PD-1 antibody）

INTERVENTIONS:
Drug: CT041 autologous CAR T-cell injection — Up to 3 times CT041 autologous CAR T-cell injection infusion
  Other Names: CAR T-cell injection
  Arms: CT041 autologous CAR T-cell injection
Drug: Physician's Choice（Paclitaxel or Irinotecan or Apatinib or Anti-PD-1 antibody） — Physician's choice of any BSC listed above
  Other Names: Best support care(BSC)
  Arms: Physician's Choice

SUMMARY:
An open, multicenter, phase Ib/II study to evaluate the efficacy, safety and pharmacokinetics of CT041 autologous CAR T-cell injection in patients with advanced gastric/ gastroesophageal junction adenocarcinoma and pancreatic cancer

DETAILED DESCRIPTION:
This study is an open, multicenter, Phase Ib/II clinical trial evaluating chimeric antigen receptor-modified autologous T cells targeting Claudin18.2 (CLDN18.2) (CT041 autologous CAR T) in subjects with CLDN18.2 expression-positive, advanced gastric/esophagogastric conjugate adenocarcinoma that has failed at least 2 prior lines therapy and advanced pancreatic cancer that has failed at least 1 prior line therapy. The purpose is to evaluate the efficacy, safety and pharmacokinetics There are two stages in the study. Phase Ib stage is dose escalation and dose expansion study, and Phase II stage is to verify the efficacy and safety of CT041 treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing to participate in a clinical trial, be informed and sign inform consent; and be willing to follow and be able to complete all trial procedures;
2. Aged 18 to 75 years;
3. Phase Ib：Patients with pathologically diagnosed advanced gastric/ gastroesophageal junction adenocarcinoma who have failed at least 2 prior lines treatment; or patients with pathologically diagnosed advanced pancreatic cancer who have failed at least 1 prior line treatment ; Phase II：Patients with pathologically diagnosed advanced gastric/ gastroesophageal junction adenocarcinoma who have failed at least 2 prior lines treatment;
4. Phase Ib：Tumor tissue samples were positive for CLDN18.2 IHC staining； Phase II：Tumor tissue samples were positive for CLDN18.2 IHC staining and HER2 expression was negative;
5. Estimated life expectancy >12 weeks;
6. According to the RECIST 1.1, there is measurable tumor lesions;
7. ECOG physical status score 0 ~ 1 at screening, within 24 hours prior to apheresis, and at baseline;
8. Sufficient venous access for mononuclear cell collection;
9. Unless otherwise specified, patients should meet the certain conditions prior to screening and pre-treatment and be allowed one week to retest if an abnormal laboratory test does not meet the criteria, and if the criteria are still not met, the screening is considered to have failed;
10. Female patients of childbearing age must undergo a serum pregnancy test at screening and prior to pretreatment and the results must be negative, and are willing to use a very effective and reliable method of contraception within 1 year after the last study treatment;
11. Men who have actively sexual intercourse with women with child-bearing potential, must agree to use barrier-based contraception if they have no vasectomy.

Exclusion Criteria:

1. Pregnant or lactating women;
2. HIV, Treponema pallidum, HCV serologically positive, EBV-DNA, CMV-DNA or 2019-ncov nucleic acid positive;
3. Any uncontrollable active infection, including but not limited to active tuberculosis, HBV infection;
4. The side effects caused by the previous treatment of the subjects did not return to CTCAE ≤1; except hair loss and other tolerable events determined by investigator;
5. Patients known to have active autoimmune diseases, including but not limited to psoriasis or rheumatoid arthritis, or other diseases requiring long-term immunosuppressive therapy;
6. Previously allergic to immunotherapy and related drugs,history of severe allergies, or allergic to components of CT041.
7. Previously received any gene-modified cell therapies(including CAR-T, TCR-T);
8. Patients have brain metastasis or symptoms of brain metastasis;
9. Patients at high risk of hemorrhage or perforation;
10. Patients requiring anticoagulant therapy;
11. Patients requiring continuous anti-platelet therapy;
12. Patients with a history of organ transplantation or awaiting organ transplantation;
13. Patients who have undergone major surgery or significant trauma within 4 weeks prior to apheresis, or who are expected to undergo major surgery during the study;
14. Presence of other serious pre-existing medical conditions that may limit patient participation in the study;
15. The investigator assessed that the patient was unable or unwilling to comply with the requirements of the study protocol;
16. The patient has a central nervous system disease sign or an abnormal neurological test result with clinical significance;
17. The patient is currently suffered from or have suffered from other incurable malignant tumors within previous 3 years, except in situ cervical cancer or skin basal cell cancer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2020-10-23 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2038-06-30 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Incidence of Treatment Related adverse events (AEs) | Up to 18 months
  Incidence of treatment related AEs, AEs of special interest and serious adverse events(SAEs).
Phase Ib: Identification of Maximum Tolerated Dose (MTD) | day1-day28
  Incidence of dose-limiting toxicities (DLTs)
Phase II: Progression-free survival (PFS), as assessed by IRC, of CT041 autologous CAR T-cell injection versus Physician's Choice | Up to 24 months
  Progression-free survival (PFS) was defined as the time from the date of randomization to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause.

SECONDARY OUTCOMES:
Phase Ib: Objective Response Rate (ORR), as assessed by Investigators | Up to 18 months
  The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.
Phase Ib: Progression-free survival (PFS), as assessed by Investigators | Up to 18 months
  Progression-free survival (PFS) was defined as the time from the date of first infusion of CT041 to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause.
Phase Ib：Overall survival (OS) | Up to 18 months
  Overall Survival (OS) was defined as the time from the date of first infusion of CT041 to the date of death due to any cause.
Phase Ib：Duration of response (DOR), as assessed by Investigators | Up to 18 months
  Duration of response (DOR) is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death.
Phase Ib：Disease control rate (DCR), as assessed by Investigators | Up to 18 months
  Disease control rate (DCR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) or Stable disease (SD) based on RECIST version 1.1.
Phase II: Overall survival (OS) of CT041 autologous CAR T-cell injection versus Physician's Choice | Up to 24 months
  Overall Survival (OS) was defined as the time from the date of randomization to the date of death due to any cause.
Progression-free survival (PFS), as assessed by Investigators, of CT041 autologous CAR T-cell injection versus Physician's Choice | Up to 24 months
  Progression-free survival (PFS) was defined as the time from the date of randomization to the earliest date of the first objective documentation of progressive disease (PD) or death due to any cause.infusion
Phase II：Objective Response Rate (ORR), as assessed by IRC and by Investigators | Up to 24 months
  The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.
Phase II: Duration of response (DOR), as assessed by IRC and by Investigators | Up to 24 months
  Duration of response (DOR) is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death.
Phase II: Disease control rate (DCR), as assessed by IRC and by Investigators | Up to 24 months
  Disease control rate (DCR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) or Stable disease (SD) based on RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Professor, Principal Investigator — Peking University Cancer Hospital & Institute; Xianjun Yu, Professor, Principal Investigator — Fudan University
Locations (24):
- China (24):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Peking University Shenzhen Hospital, Shenzhen, Guangzhou
  - Harbin medical university Affiliated Cancer Hospital, Harbin, Heilongjia
  - Henan Tumor Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science & Technology, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Ruijin Hospital, affiliated to Shanghai Jiaotong University, school of medicine, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Shanghai Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qi C, Liu C, Peng Z, Zhang Y, Wei J, Qiu W, Zhang X, Pan H, Niu Z, Qiu M, Qin Y, Fang W, Ye F, Li N, Liu T, Liu A, Zhang X, Hu C, Zhang J, Cui J, Lin X, Wang S, Zhang J, Lin T, Qu X, Yuan X, Gong J, Li J, Gao W, Gai L, Wang Y, Yuan D, Li Z, Shen L. Claudin-18 isoform 2-specific CAR T-cell therapy (satri-cel) versus treatment of physician's choice for previously treated advanced gastric or gastro-oesophageal junction cancer (CT041-ST-01): a randomised, open-label, phase 2 trial. Lancet. 2025 Jun 7;405(10494):2049-2060. doi: 10.1016/S0140-6736(25)00860-8. Epub 2025 May 31. PMID 40460847
- [Derived] Qi C, Zhang P, Liu C, Zhang J, Zhou J, Yuan J, Liu D, Zhang M, Gong J, Wang X, Li J, Zhang X, Li N, Peng X, Liu Z, Yuan D, Baffa R, Wang Y, Shen L. Safety and Efficacy of CT041 in Patients With Refractory Metastatic Pancreatic Cancer: A Pooled Analysis of Two Early-Phase Trials. J Clin Oncol. 2024 Jul 20;42(21):2565-2577. doi: 10.1200/JCO.23.02314. Epub 2024 May 24. PMID 38788174
- [Derived] Qi C, Xie T, Zhou J, Wang X, Gong J, Zhang X, Li J, Yuan J, Liu C, Shen L. CT041 CAR T cell therapy for Claudin18.2-positive metastatic pancreatic cancer. J Hematol Oncol. 2023 Sep 9;16(1):102. doi: 10.1186/s13045-023-01491-9. PMID 37689733